CLINICAL TRIAL: NCT04993287
Title: The Cascade Feasibility Pilot (HF): Improving Care Processes for Heart Failure Patients Using Continuous Remote Patient Monitoring and a Cascading Alert System
Brief Title: The Cascade Feasibility Pilot (HF) Phase 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Nirav Shah, Medical Director of Quality Innovation and Clinical Practice Analytics, Program Director of Outcomes Research for Quality and Transformation, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EH20-288 Cascade HF
Record Dates: First submitted 2021-07-16; First posted 2021-08-06 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pilot (Experimental): 39 eligible HF patients
  Interventions: Other: Non-invasive continuous remote monitoring with structured escalation pathway; Other: Affective Analysis of Participant Response to Continuous Remote Patient Monitoring

INTERVENTIONS:
Other: Non-invasive continuous remote monitoring with structured escalation pathway — Continuous patient monitoring through non-invasive biosensors coupled with machine learning algorithms, with a structured escalation and communication pathway for home health providers and HF care team
Other: Affective Analysis of Participant Response to Continuous Remote Patient Monitoring — Surveys and interviews with enrolled participants

SUMMARY:
The study proposal is to deploy a wearable solution that predicts physiological perturbation comparable to invasive devices and to perform continuous remote patient monitoring; this will be connected to a structured, cascading, escalation pathway involving home health nurses, advanced practitioner providers, and heart failure specialists, and has the potential to transform heart failure management in the post-discharge period, where patients are the most vulnerable for readmission. This feasibility study will contribute to the understanding of post-discharge heart failure continuous remote patient monitoring, promote patient self-care, and has the potential of improving patient outcomes.

DETAILED DESCRIPTION:
Heart failure is a leading cause of hospital readmission. It results in significant mortality, morbidity, and health care utilization. Effective continuous remote patient monitoring (CRPM) can reduce readmissions, but it has only been realized via invasive monitoring. The study will focus on non-invasive heart failure CRPM through a structured cascading and escalating alert system. In this feasibility study, the study team will use a wearable biosensor and collect ambulatory physiological data that are analyzed by machine learning algorithms, potentially identifying physiological perturbation in heart failure patients. Alerts from this algorithm may be cascaded with other patient status data to inform management by the home health team via a structured protocol. The escalation pathway will engage home health, advanced practitioner providers, and heart failure specialists. In the first aim, the study team will perform a soft launch on five patients with an extensive evaluation to assess feasibility for the pilot trial. In aim 2, the study team will implement the feasibility pilot study. In aim 2a, the study team will conduct surveys and semi-structured interviews with both providers and patients. The surveys and interviews will be applied at three time points (initiation, maintenance, and post-study) to evaluate perceptions, acceptance, and experience of this CRPM solution. In aim 2b, the investigators will leverage temporal data mining, feature extraction, and patient clustering methods to identify valid patterns associated with the pathophysiological events of interest, using continuous physiological data, patient reports, and electronic health record data. The study team will also compare outcome and process measures from our pilot study to a retrospective cohort matched for key demographics and disease severity. This feasibility study will provide key learning for a larger efficacy clinical trial to evaluate if this non-invasive telemonitoring solution tied to structured patient management via cascading and escalating alert pathways can improve outcomes and reduce heart failure readmission.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an inpatient at Evanston Hospital
* Patient is followed by the heart failure service team after discharge
* Patient has a history of heart failure
* Patient received at least one dose of IV diuretic at index hospitalization
* Symptoms corresponding to NYHA function class II-IV
* Patient has heart failure with reduced left ventricular ejection fraction (LVEF)<40%, or HF with mid-ranged ejection fraction (LVEF 40-50%), or HF with preserved ejection fraction (LVEF≥50%)
* Patient is in the top 50% risk of readmission across NorthShore University HealthSystem's CAPE 30-day readmission model
* Patient is at least 18 years of age
* Patient is fluent in English
* Patient agrees to protocol-required procedures

Exclusion Criteria:

* Patient has cognitive or physical limitations that, in the investigator's opinion, limit the patient's ability to maintain patch device and phone
* Patient has visual impairments
* Patient has an allergy to hydrocolloid adhesives
* Patient has present skin damage preventing them from wearing a study device
* Patient has renal dysfunction requiring dialysis
* Patient has CardioMEMS
* Pregnancy
* Patient receiving hospice care

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nirav S Shah, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem Evanston Hospital, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study approached a total of 61 potential participants that signed that consent forms. Out of which 39 completed the study, 16 were screen failed and 6 withdrew the consent.
  15 providers participated in the study
Groups:
- 15 HF Providers Were Included in the Study: HF providers who were part of advanced cardiology services were included in the study
  Non-invasive continuous remote monitoring with structured escalation pathway: Continuous patient monitoring through non-invasive biosensors coupled with machine learning algorithms, with a structured escalation and communication pathway for home health providers and HF care team
Period: Overall Study
Arm/Group | Pilot | 15 HF Providers Were Included in the Study
Started | 39 | 15
Completed | 39 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics and/or adverse events were not collected from clinical team staff.
Groups:
- Pilot: 39 eligible HF patients and 15 HF providers
  Non-invasive continuous remote monitoring with structured escalation pathway: Continuous patient monitoring through non-invasive biosensors coupled with machine learning algorithms, with a structured escalation and communication pathway for home health providers and HF care team
  Affective Analysis of Participant Response to Continuous Remote Patient Monitoring: Surveys and interviews with enrolled participants
  Baseline characteristics were not collected for HF proivders
Arm/Group | Pilot
Number analyzed (Participants) | 39
Age, Customized [Median (Inter-Quartile Range); unit: Years] | 75 [68 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 4
  Asian | 4
  Caucasian | 24
  Hispanic | 1
  Other | 6
Smoking [Count of Participants; unit: Participants]
  Current | 2
  Former | 19
  Never | 18
Comorbidities [Count of Participants; unit: Participants]
  Diabetes Mellitus | 17
  Hypertension | 29
  CKD | 23
  COPD | 9
  AFIB | 17
  Obesity (BMI) | 20
  Depression | 12
  Anxiety | 13
  Myocardial infarction | 4
  Implantable Defibrillator | 7
  Cardioversion/Cardiac Resynchronization Therapy | 4
Heart Failure Severity [Count of Participants; unit: Participants] — Heart failure severity is described based on New York Heart Association (NYHA) Classification and type of heart failure:
  Class I - No physical activity limitation. Ordinary activity doesn't cause fatigue, palpitations, or breathlessness.
  Class II - Slight limitation. Comfortable at rest, but ordinary activity causes fatigue, palpitations, breathlessness, or chest pain.
  Class III - Marked limitation. Comfortable at rest, but less than ordinary activity triggers symptoms.
  Class IV - Symptoms at rest. Any activity worsens discomfort.
  Higher class indicates greater severity.
  Participants
    New York Heart Association Class II | 4
    New York Heart Association Class III | 30
    New York Heart Association Class IV | 5
    Diastolic Heart Failure | 17
    Systolic Heart Failure | 6
    Systolic and Diastolic Heart Failure | 15
    Unspecified Type of Heart Failure | 1
    Heart Catherization in Index Stay | 12
Ejection Fraction [Median (Inter-Quartile Range); unit: Percentage] — Ejection fraction (EF) is a measurement, expressed as a percentage, of how much blood the left ventricle pumps out with each contraction. A normal heart's ejection fraction is between 55 and 70 percent.
  Percentage | 52 [33.4 to 64]
Ejection Fraction Type [Count of Participants; unit: Participants] — Heart failure with preserved ejection fraction (HFpEF): Patients with ejection fraction of greater than or equal to 50% Heart failure mid-range ejection fraction (HFmrEF): Patients with ejection fraction ejection fraction between 41% and 49% Heart failure reduced ejection fraction (HFrEF): Patients with ejection fraction of less than or equal to 39%
  Participants
    Heart failure with preserved ejection fraction (Ejection Fraction of greater than or equal to 50%) | 21
    Heart failure with mid-range ejection fraction (Ejection Fraction of 41% to 49%) | 4
    Heart failure with reduced ejection fraction (Ejection Fraction of less than 39%) | 14
Clinical Analytics Prediction Engine (CAPE) Readmission Risk Score [Median (Inter-Quartile Range); unit: Percentage] — Clinical Analytics Prediction Engine (CAPE) is a custom 30-day readmission risk prediction model that detects patient deterioration. The score is presented in percentage (0-100%). Higher percentage score represents higher risk of readmission.
  Percentage | 18 [13.5 to 24]
Insurance Type [Count of Participants; unit: Participants]
  Commercial | 10
  Government | 0
  Medicaid | 2
  Medicare | 25
Discharge Medications [Count of Participants; unit: Participants]
  Digoxin | 6
  Loop diuretics | 36
  ACE/ARB-Antihypertensive medications | 11
  Beta blockers | 29
  Aldosterone Agonist - Spironolactone | 24

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: Enrollment rate for entire patient cohort
Time Frame: Through study completion, an average 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot
Number analyzed (Participants) | 39
Participants | 39

2. Primary Outcome: Adherence Rate
Description: Patient adherence to electronic patient reported outcomes
Time Frame: Through study completion, an average of one year
Population: Number of patients completed at least 80% of the electronic patient reported outcomes survey
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot
Number analyzed (Participants) | 39
Participants | 27

3. Secondary Outcome: Documented Diuretic Escalation
Description: Number of patients on escalated diuretics dosage by the clinical care team during monitoring period
Time Frame: 30 days from patient discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot
Number analyzed (Participants) | 39
Participants | 17

4. Secondary Outcome: 30-day Readmission Rate
Description: 30-day readmission rate from the day of discharge
Time Frame: 30 days from patient discharge date
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot
Number analyzed (Participants) | 39
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 30 days after discharge for the enrolled HF patients. HF providers were not monitored/assessed for adverse events.
Groups:
- Pilot - 39 Eligible HF Patients: 39 eligible HF patients
  Non-invasive continuous remote monitoring with structured escalation pathway: Continuous patient monitoring through non-invasive biosensors coupled with machine learning algorithms, with a structured escalation and communication pathway for home health providers and HF care team
  Affective Analysis of Participant Response to Continuous Remote Patient Monitoring: Surveys and interviews with enrolled participants
Arm/Group | Pilot - 39 Eligible HF Patients
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT04993287/Prot_000.pdf